CLINICAL TRIAL: NCT05131126
Title: Influence of an Anterior Latarjet-type Abutment Operation on Scapular Dyskinesia and the Muscular Stabilization Mechanisms of the Scapula (DyScapLat)
Acronym: DyScapLat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-A02449-46
Record Dates: First submitted 2021-11-10; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Latarjet; Scapular Dyskinesis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient requiring anterior abutment surgery by Latarjet method (Experimental)
  Interventions: Procedure: Latarjet method; Other: Different arms exercices
- Healthy volunteers (Active Comparator)
  Interventions: Other: Different arms exercices

INTERVENTIONS:
Procedure: Latarjet method — This operation consists of fixing a bone graft
  Arms: Patient requiring anterior abutment surgery by Latarjet method
Other: Different arms exercices — Perform 5 elevation movements in each of the elevation planes (sagittal, scapular and coronal) with the right and left arms
  * Perform 5 circumduction movements with the right and left arms
  * Maintain a weight of 1kg twice for 5 seconds with the arms at 90 ° of elevation.

SUMMARY:
The aim of this study is to assess the influence of anterior abutment surgery using the Latarjet method on the kinematics of the scapula. The sub-objectives will be to show that Latarjet-type surgery does not lead to scapular dyskinesia and modification of muscle activity compared to a control group that has not undergone an operation.

ELIGIBILITY:
Inclusion Criteria:

* Patient Group:

  * Male between 18 and 40 years-old
  * Practice a regular sports activity before the injury (s) requiring surgery
  * Present the clinical criteria leading to anterior abutment surgery using the Latarjet method
  * Surgery performed by surgeons from the Jean-Mermoz Private Hospital (69008 Lyon)
  * Have followed a post-surgery self-rehabilitation program

Control group:

* Male between 18 and 40 years-old
* Practice a regular sports activity

Both group:

oPatient having signed an informed consent o Subject affiliated or beneficiary of a social security scheme

Exclusion Criteria:

Patient group:

* Have another shoulder pathology on the side of the operated limb or on the contralateral side
* Present a constitutional hyper laxity
* Have stiffness or recurrence of dislocation of the shoulder post-surgery
* Have a body mass index greater than 30 kg / m² (to ensure sufficient accuracy to measure the movements of the scapula)
* Wear a pacemaker or any other metal device (e.g. patch with metal material)
* Present a contraindication to the use of measuring devices (intolerance to a weak electromagnetic field)

Control group:

* Present during the study or have presented in the past any musculoskeletal pathology in the right or left shoulder (WOSI or WORC score greater than 250).
* Have a body mass index greater than 30 kg / m² (to ensure sufficient accuracy to measure the movements of the scapula)
* Wear a pacemaker or any other metal device (e.g. patch with metal material)
* Present a contraindication to the use of measuring devices (intolerance to a weak electromagnetic field)

Both group :

o Protected subject: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05-22 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2023-05-22 (Estimated)

PRIMARY OUTCOMES:
Difference in position of the scapula (tilt, rotation and bell) between the pre and post-test measured in the control group | 4 months
  For electromyographic analysis, the signals will be filtered, smoothed and normalized to obtain a percentage of activation relative to that measured during submaximal voluntary contractions.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital privé Jean Mermoz, Lyon, France